CLINICAL TRIAL: NCT04432064
Title: Temporal Interference Neurostimulation and Addiction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemic restrictions delayed data collection and led to loss of funding.
Sponsor: Indiana University (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Joshua Brown, PHD, Professor, Psychological and Brain Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1904451651
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Nicotine Use Disorder; Substance Use Disorders
Keywords: Nicotine Addiction; Non-invasive deep brain stimulation; Substance Use Disorders
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: One group of 20 participants will receive active TI-NDBS and another group of 20 participants will receive sham TI-NDBS. A third group of 20 participants will receive traditional transcranial direct current stimulation (tDCS).
Who Masked: Participant
Masking Description: This will be single-blind masking as the experimenter will need to know which intervention to run on the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Phase 3 Active TI-NDBS (Experimental): Participants assigned to this condition will receive active temporal interference non-invasive deep brain stimulation. Participants will receive stimulation for 60 minutes on one day.
  Interventions: Device: Active TI-NDBS
- Phase 3 Sham TI-NDBS (Sham Comparator): Participants assigned to this condition will receive sham temporal interference non-invasive deep brain stimulation, in which they will have electrodes attached to the scalp but the device is only turned on for a few seconds.
  Interventions: Other: Sham TI-NDBS
- Phase 4 Traditional tDCS (Active Comparator): Participants assigned to this condition will receive traditional transcranial direct current stimulation for 60 minutes for 5 days.
  Interventions: Device: tDCS
- Phase 4 TI-NDBS (Experimental): Participants assigned to this condition will receive active temporal interference non-invasive deep brain stimulation for 60 minutes for 5 days and will be compared to sham stimulation and tDCS.
  Interventions: Device: Active TI-NDBS
- Phase 4 Sham stimulation (Sham Comparator): Participants assigned to this condition will receive sham temporal interference non-invasive deep brain stimulation, in which they will have electrodes attached to the scalp but the device is only turned on for a few seconds. Participants will be in the scanner for 60 minutes for 5 days. This will be used as the control condition and compared with TI-NDBS and tDCS.
  Interventions: Other: Sham TI-NDBS

INTERVENTIONS:
Device: Active TI-NDBS — In the active TI-NDBS condition, subjects will receive stimulation for 60 minutes applied to the brain through scalp electrodes. There will be a maximum of 2 mA per electrode pair and no single region will receive more than 2 mA because the currents will be administered to distinct regions. At the beginning of each stimulation period, the current will increase slowly at a constant rate for 30 seconds until it reaches the appropriate intensity. At the end of the stimulation, the current will decrease slowly for 30 seconds until it reaches zero.
  Other Names: Temporal Interference Non-invasive Deep Brain Stimulation
  Arms: Phase 3 Active TI-NDBS; Phase 4 TI-NDBS
Other: Sham TI-NDBS — This is the control condition in which participants will receive sham stimulation for 60 minutes.
  Arms: Phase 3 Sham TI-NDBS; Phase 4 Sham stimulation
Device: tDCS — This is a well established method of brain stimulation and will be used to compare against the efficacy of TI-NDBS in the reduction of nicotine craving and inhalation. Participants will receive stimulation for 60 minutes.
  Arms: Phase 4 Traditional tDCS

SUMMARY:
This project aims to develop a line of research using new non-invasive neurostimulation technology to treat adults with opioid use disorders (OUDs). In the short term, the investigators aim to identify novel target brain regions for neurostimulation treatment and characterize their effects behaviorally and neurally. In the longer term, investigators aim to use these preliminary data to justify NIH sponsored clinical trials to apply transcranial direct current stimulation and non-invasive deep brain stimulation to these areas to partially or completely disrupt addiction.

DETAILED DESCRIPTION:
The investigators hypothesize that temporal interference non-invasive deep brain stimulation (TI-NDBS) will be well tolerated and effective at manipulating brain activity and reducing drug cravings. The investigators will investigate whether stimulation with a mild current from temporal interference non-invasive deep brain stimulation (TI-NDBS) to the Anterior Cingulate Cortex (ACC), the anterior insula (AI), or the nucleus accumbens (NAcc) will reduce nicotine craving and seeking. The TI-NDBS is similar to the traditional transcranial direct current stimulation (tDCS), a method approved for use in a number of other studies. Other studies have shown there have been some effects of reducing craving with tDCS, however, tDCS cannot stimulate structures such as the ACC very effectively because tDCS cannot stimulate deeper brain regions. Thus, the Specific Aim ultimately will compare TI-NDBS with tDCS and sham stimulation. The study is broken up into four phases. The first two will involve device feasibility and identifying the best locations for the electrodes to be placed. In the third phase, the investigators will compare TI-NDBS with sham stimulation. In the fourth phase, the investigators will compare TI-NDBS with sham stimulation and with tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 50, must have at least 6th grade education, and the ability to speak and read English, must smoke at least 3/4 of a pack of cigarettes per day, must have phone with internet access.

Exclusion Criteria:

* if they are on psychotropic medications for ADHD, other mental illness or medication for cancer, epilepsy (i.e. individuals with any history of seizure disorder), migraines, or other neurological syndromes, or AIDs (which can cause cognitive deficits (Watkins & Treisman, 2015), history of head trauma, history of cognitive impairments, metal implants in the head or under the scalp, personal experiences consistent with symptoms of psychosis (i.e. mind or body being secretly controlled, special powers, seeing or hearing things that aren't really there).
* Subjects will be excluded if they do not meet fMRI safety screening criteria (i.e. metal implants in their body, tattoo on head or neck, permanent jewelry, etc.) or if a participant uses an IUD for birth control they will be excluded unless the subject can document the model of the IUD and we can verify its safety for the MRI environment. Pregnancy should be self-reported, and a pregnancy test will not be administered. Participants must also weigh less than 440 lbs.
* History of holes bored into skull or known fissures in cranial bones
* Presence of pacemakers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share anonymized participant data upon request. Beyond that, we will report anonymized data publicly in aggregate.

REFERENCES:
- [Background] Fregni F, Liguori P, Fecteau S, Nitsche MA, Pascual-Leone A, Boggio PS. Cortical stimulation of the prefrontal cortex with transcranial direct current stimulation reduces cue-provoked smoking craving: a randomized, sham-controlled study. J Clin Psychiatry. 2008 Jan;69(1):32-40. doi: 10.4088/jcp.v69n0105. PMID 18312035
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- [Background] Fecteau S, Agosta S, Hone-Blanchet A, Fregni F, Boggio P, Ciraulo D, Pascual-Leone A. Modulation of smoking and decision-making behaviors with transcranial direct current stimulation in tobacco smokers: a preliminary study. Drug Alcohol Depend. 2014 Jul 1;140:78-84. doi: 10.1016/j.drugalcdep.2014.03.036. Epub 2014 Apr 16. PMID 24814566
- [Background] Hulvershorn LA, Hummer TA, Fukunaga R, Leibenluft E, Finn P, Cyders MA, Anand A, Overhage L, Dir A, Brown J. Neural activation during risky decision-making in youth at high risk for substance use disorders. Psychiatry Res. 2015 Aug 30;233(2):102-11. doi: 10.1016/j.pscychresns.2015.05.007. Epub 2015 May 21. PMID 26071624
- [Background] Wing VC, Barr MS, Wass CE, Lipsman N, Lozano AM, Daskalakis ZJ, George TP. Brain stimulation methods to treat tobacco addiction. Brain Stimul. 2013 May;6(3):221-30. doi: 10.1016/j.brs.2012.06.008. Epub 2012 Jul 9. PMID 22809824
- [Background] Velez de Mendizabal N, Jones DR, Jahn A, Bies RR, Brown JW. Nicotine and cotinine exposure from electronic cigarettes: a population approach. Clin Pharmacokinet. 2015 Jun;54(6):615-26. doi: 10.1007/s40262-014-0221-7. PMID 25503588
- [Background] Naqvi NH, Rudrauf D, Damasio H, Bechara A. Damage to the insula disrupts addiction to cigarette smoking. Science. 2007 Jan 26;315(5811):531-4. doi: 10.1126/science.1135926. PMID 17255515
- [Background] Naqvi NH, Gaznick N, Tranel D, Bechara A. The insula: a critical neural substrate for craving and drug seeking under conflict and risk. Ann N Y Acad Sci. 2014 May;1316:53-70. doi: 10.1111/nyas.12415. Epub 2014 Apr 1. PMID 24690001
- [Background] Muller UJ, Sturm V, Voges J, Heinze HJ, Galazky I, Heldmann M, Scheich H, Bogerts B. Successful treatment of chronic resistant alcoholism by deep brain stimulation of nucleus accumbens: first experience with three cases. Pharmacopsychiatry. 2009 Nov;42(6):288-91. doi: 10.1055/s-0029-1233489. Epub 2009 Nov 18. No abstract available. PMID 19924591
- [Background] Craig AD. How do you feel? Interoception: the sense of the physiological condition of the body. Nat Rev Neurosci. 2002 Aug;3(8):655-66. doi: 10.1038/nrn894. PMID 12154366

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 3 Active TI-NDBS | Phase 3 Sham TI-NDBS | Phase 4 Traditional tDCS | Phase 4 TI-NDBS | Phase 4 Sham Stimulation
Started | 10 | 0 (Not started) | 0 (not started) | 0 (not started) | 0 (not started)
Completed | 5 | 0 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: COVID delays and lack of funding
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 3 Active TI-NDBS | Phase 3 Sham TI-NDBS | Phase 4 Traditional tDCS | Phase 4 TI-NDBS | Phase 4 Sham Stimulation | Total
Number analyzed (Participants) | 10 | 0 | 0 | 0 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 0 | 0 | 0 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  |  |  |  | 6
  Male | 4 |  |  |  |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  |  | 0
  Not Hispanic or Latino | 10 |  |  |  |  | 10
  Unknown or Not Reported | 0 |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  |  | 0
  Asian | 0 |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  | 0
  Black or African American | 0 |  |  |  |  | 0
  White | 10 |  |  |  |  | 10
  More than one race | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 |  |  |  |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Nicotine Craving
Description: The investigators predict that TI-NDBS will outperform sham stimulation at an overall change in smoking and cigarette craving, which in turn will outperform sham stimulation. The investigators will sum the total inhaled nicotine vapor volume in liters over the 60 minute session and perform pairwise t-tests to determine if total drug intake is lower with TI-NDBS vs tDCS. Also, the investigators will average the self reported craving levels on a Likert scale across each subject during the 60 minute session, and the investigators will perform pairwise tests to determine if stimulation lowers self reported craving. **The Likert scale is 0-10, where 10 is maximum craving. The units are units on a scale.** **The outcome measure is computed by taking the pre-stimulation craving and subtracting the post-stimulation craving. Positive numbers indicate the degree to which the self-reported craving was reduced after the stimulation relative to before stimulation**
Time Frame: Each subject was asked to report their craving during the day of the session, before and after the stimulation. Approximately one hour elapsed between before and after nicotine craving measurements. The session was carried out during the daytime.
Population: Note the results here cannot be interpreted meaningfully as we were unable to run the control group, so there is no valid comparison.
Measure: Mean (Standard Deviation); unit: reduction in nicotine craving on 10-pt
Arm/Group | Phase 3 Active TI-NDBS
Number analyzed (Participants) | 5
reduction in nicotine craving on 10-pt | 4.25 (1.71)

ADVERSE EVENTS:
Time Frame: The total duration of collecting information about adverse events across subjects was 1 year, 5 months. Each individual subject was monitored for adverse events over a one day period.
Arm/Group | Phase 3 Active TI-NDBS
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 3 Active TI-NDBS (N=10)
Unpleasant sensation (Skin and subcutaneous tissue disorders) | 1 (1) — Subject experienced unpleasant sensation on the scalp which required terminating the session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04432064/Prot_SAP_000.pdf